CLINICAL TRIAL: NCT02269709
Title: Noninvasive Detection of Liver Injury Immediately Following the Fontan Operation: the Role of Ultrasound-Based Elastography
Brief Title: Stage 3 Fontan Operation Liver Ultrasound Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Frank Dipaola, Principal Investigator, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00090329
Record Dates: First submitted 2014-10-15; First posted 2014-10-21 (Estimated); Results first posted 2017-08-16 (Actual); Last update posted 2018-01-12 (Actual); Status verified 2017-11

CONDITIONS: Fontan Operation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ARFI Ultrasound (Experimental): This study uses ultrasound scanning with acoustic radiation force impulse shear wave velocity imaging to measure pediatric liver fibrosis. Patients will be children who have had the Fontan operation. This is a non-invasive scan that uses sound waves to create images.
  Interventions: Device: ARFI Ultrasound

INTERVENTIONS:
Device: ARFI Ultrasound — This research scan uses acoustic radiation force impulse (ARFI) shear wave velocity imaging (SVI). This is a new ultrasound technology in which unique sound waves create the images/pictures of the liver beng examined/scanned. This ultrasound scan will take approximately 10 minutes to complete.

SUMMARY:
The purpose of this study is to compare the liver stiffness, which can be caused by congestion and fibrosis in pediatric patients before and after a Fontan heart operation.

A new form of ultrasound elastography (Acoustic Radiation Force Impulse, or ARFI) will measure liver stiffness.

DETAILED DESCRIPTION:
The Fontan repair for single ventricle congenital heart lesions consists of three stages. This surgery has enable pediatric patients who have the repair to live into adulthood.

Stage 3 of the surgery introduces immediate congestion of blood in the liver by increasing central venous pressure (CVP). CVP is the blood pressure within the vena cava, a major blood vessel in the body.

Many patients later develop progressive liver fibrosis (stiffness) possibly as a result of increased blood pressure. Liver stiffness is increased both by congestion and fibrosis.

Liver fibrosis has significant health risks and may complicate the patient's future healthcare.

There are no established, noninvasive means of detecting the liver fibrosis until it becomes severe. Acoustic radiation force impulse (ARFI) elastography, an ultrasound technique, can measure the stiffness of the liver safely from outside the body.

The investigators hypothesize that liver stiffness will be increased by stage 3 of the Fontan operation due to onset of liver congestion.

Using ARFI, the investigators will measure liver stiffness before and immediately after stage 3 of the Fontan operation, when congestion of blood is likely the only contributor to any change in liver stiffness.

The investigators will follow the trend of liver stiffness at six months by repeating the ARFI imaging.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients ages 0-17
* Patients presenting to the University of Michigan for evaluation just before undergoing stage 3 of the Fontan operation

Exclusion Criteria:

* Patients over the age of 17
* Patients who have chronic liver disease (elevation of ALT, AST, or Bilirubin greater than two times the upper limits of normal >4 weeks)
* Patients who have evidence of liver enlargement or nodularity on prior ultrasound imaging
* Patients who have a history of portal vein or hepatic vein thrombosis
* Patients (parents) who are unwilling to read and sign the informed consent document

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2014-11; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank W DiPaola, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ARFI Ultrasound: Subjects were pediatric patients who had undergone a repair of a heart defect, called a Fontan operation. Patients underwent an ultrasound before and after the Fontan operation.
  The ultrasound scan used acoustic radiation force impulse (ARFI) shear wave velocity imaging (SVI). This is a non-invasive scan that uses sound waves to create images of the liver and measure its stiffness.
Period: Time of Enrollment
Arm/Group | ARFI Ultrasound
Started | 21
Completed (Three patients withdrew before the start of the study.) | 18
Not Completed | 3
Not completed — Withdrawal by Subject | 3
Period: Follow-up #1 (24-72 Hours Post-surgery)
Arm/Group | ARFI Ultrasound
Started | 18
Completed | 17
Not Completed | 1
Not completed — Lost to Follow-up | 1
Period: Prior to Hospital Discharge
Arm/Group | ARFI Ultrasound
Started | 17
Completed | 17
Not Completed | 0
Period: Six Month Follow-up
Arm/Group | ARFI Ultrasound
Started | 17
Completed | 5
Not Completed | 12
Not completed — Lost to Follow-up | 12

BASELINE CHARACTERISTICS:
Groups:
- ARFI Ultrasound: Subjects were pediatric patients who had undergone a Fontan operation. Subjects underwent an ultrasound before and after the Fontan operation. The ultrasound scan used acoustic radiation force impulse (ARFI) shear wave velocity imaging (SVI). This is a non-invasive scan that uses sound waves to create images of the liver and measure the stiffness of the tissue.
Arm/Group | ARFI Ultrasound
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: Months] | 33.5 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 12
Age by Sex [Mean (Full Range); unit: Months] — Population: The age of each gender group (males and females) is compared.
  Months
    Age of Male Subjects: number analyzed (Participants) | 12
    Age of Male Subjects | 34 [18 to 52]
    Age of Female Subjects: number analyzed (Participants) | 6
    Age of Female Subjects | 33 [24 to 47]

OUTCOME MEASURES:

1. Primary Outcome: Shear Wave Speed (Liver Stiffness)
Description: ARFI shear wave speed measurements were done on the right lobe of the liver. Measurement units are m/s (meters per second). A total of 8 measurements were performed on each subject at each time point.The 8 values were performed on each subject and averaged.
Time Frame: 0-6 months
Population: As shown in the participant flow, data was not captured for follow up time points 1 and 2 for 1 participant. At time point 3 data is only available for 5 participants.
Measure: Mean (Standard Deviation); unit: meters per second
Groups:
- ARFI Ultrasound: Subjects underwent an ultrasound scan before and after the Fontan operation.
Arm/Group | ARFI Ultrasound
Number analyzed (Participants) | 18
meters per second
  Liver Stiffness at baseline | 1.18 (0.29)
  Liver Stiffness follow-up tim1 (24-72 hours later): number analyzed (Participants) | 17
  Liver Stiffness follow-up tim1 (24-72 hours later) | 2.28 (0.31)
  Liver Stiffness follow-up time 2 (7 days later): number analyzed (Participants) | 17
  Liver Stiffness follow-up time 2 (7 days later) | 2.22 (0.38)
  Liver stiffness follow-up time 3 (6 months): number analyzed (Participants) | 5
  Liver stiffness follow-up time 3 (6 months) | 2.08 (0.24)
Statistical Analysis 1: Comparison: ARFI Ultrasound; Comparison of Baseline and Follow-up #1; Test type: Other — Changes in mean liver shear wave speed (SWS) between time points were assessed using a mixed-effect model with post hoc Tukey correction; p < 0.0001, Mixed Models Analysis
Statistical Analysis 2: Comparison: ARFI Ultrasound; Comparison of Baseline vs. Follow up #2; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed Models Analysis
Statistical Analysis 3: Comparison: ARFI Ultrasound; Comparison of Baseline vs. Follow-up #3; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed Models Analysis

2. Secondary Outcome: IVC Pressure
Description: Blood pressure in the IVC, the interior vena cava, was measured from a central line placed for patient care.
Time Frame: Baseline and Follow Up Number 1 (approximately 24 -72 hours later)
Population: Subjects who had undergone the Fontan operation and who had a central line placed. Blood pressure values were obtained from chart review.
Measure: Mean (Standard Error); unit: mmHg
Groups:
- ARFI Ultrasound: Subjects underwent an ultrasound scan before and after the Fontan operation. The blood pressure in the IVC (interior vena cava) was measured.
Arm/Group | ARFI Ultrasound
Number analyzed (Participants) | 9
mmHg
  IVC pressure before Fontan operation | 7.2 (2.6)
  IVC pressure after Fontan operation (24-72 hours) | 16.44 (3.3)
Statistical Analysis 1: Comparison: ARFI Ultrasound; Test type: Other — Mean IVC pressures from different time points were compared using the Wilcoxon signed-rank test; p < 0.05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Patients were followed for adverse events through their last hospital visit which was up to 6 months at the latest.
Arm/Group | ARFI Ultrasound
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

LIMITATIONS AND CAVEATS:
The study is limited by the small sample size and the limited capture of follow-up Ultrasound Shear Wave Elastography data at the 6 month time point. Most patients who underwent Fontan operations received follow-up care closer to home.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes